CLINICAL TRIAL: NCT01424852
Title: Early Administration of Bifidobacterium Lactis BB-12 and the Caries Occurence of Children a 4 Years of Age
Brief Title: Does Administration of Probiotics During Infancy Increase the Caries Risk of a Child
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Too few of the invited subjects wanted to participate
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Eva Soderling, Adjunct Professor, University of Turku
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Probiotics study7.4.2011
Record Dates: First submitted 2011-08-26; First posted 2011-08-29 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Dental Caries
Keywords: Probiotics; Caries; Oral flora
MeSH Terms: conditions — Dental Caries | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotics in milk formula (Active Comparator): B. lactis BB-12 and L. rhamnosus GG delivered in milk formula during the first year of infancy
  Interventions: Dietary Supplement: Probiotics in infant milk formula
- Control milk formula (Placebo Comparator): The children received milk formula with no probiotics
  Interventions: Dietary Supplement: Probiotics in infant milk formula

INTERVENTIONS:
Dietary Supplement: Probiotics in infant milk formula — Probiotic infgant milk formula administered during the forst year of life
  Other Names: B.lactis BB12 and L.rhamnosus GG in milk formula

SUMMARY:
Aim: to examine caries occurrence in children who ten years ago received a mixture of probiotics during infancy.

Hypothesis: the administration of probiotics during infancy has no effect on future dental health.

ELIGIBILITY:
Inclusion Criteria:

* Child participated in the probiotic milk intervention study in early 2000
* Child lives now within 100 km from Turku

Exclusion Criteria:

* Child has a chronic illness affecting dental health
* Child lives now outside 100 km from Turku

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Caries occurence | 10 years

SECONDARY OUTCOMES:
Oral microbial colonization | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Erika M Isolauri, Professor, Study Director — University of Turku
Locations (1):
- University of Turku, Turku, Finland, Finland